CLINICAL TRIAL: NCT01178372
Title: Secondary Prophylaxis of Hepatic Encephalopathy in Cirrhosis: An Open Label, Randomized Controlled Trial of Lactulose, Probiotics and No-therapy
Brief Title: Secondary Prophylaxis of Hepatic Encephalopathy in Cirrhosis
Acronym: HE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Govind Ballabh Pant Hospital (Other Government)
Other Study IDs: PS002
Record Dates: First submitted 2010-08-09; First posted 2010-08-10 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2009-09

CONDITIONS: Hepatic Encephalopathy
Keywords: hepatic encephalopathy; lactulose; probiotics
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Lactulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lactulose (Active Comparator): will receive 30-60 ml of lactulose in 2 or 3 divided doses so that patient passed 2-3 semisoft stools per day
  Interventions: Drug: Lactulose
- probiotics (Active Comparator)
  Interventions: Drug: Probiotics(VSL#3)

INTERVENTIONS:
Drug: Lactulose — will receive 30-60 ml of lactulose in 2 or 3 divided doses so that patient passed 2-3 semisoft stools per day
  Arms: lactulose
Drug: Probiotics(VSL#3) — will receive VSL#3 (110 billion CFU)three times a day
  Arms: probiotics

SUMMARY:
Hepatic encephalopathy (HE), a challenging complication of advanced liver disease, occurs in approximately 30-45% of patients with cirrhosis. The treatment of choice is non-absorbable disaccharides, such as lactulose and lactitol.Probiotics are effective in the treatment of minimal hepatic encephalopathy which precipitates hepatic encephalopathy. The investigators will assess the effects of lactulose and probiotics for the prevention of recurrence of HE (secondary prophylaxis) in patients after the recovery of an episode of overt hepatic encephalopathy.

DETAILED DESCRIPTION:
Hepatic encephalopathy, a challenging complication of advanced liver disease, occurs in approximately 30-45% of patients with cirrhosis and 10-50% of patients with transjugular intrahepatic portosystemic shunt.Although the occurrence of episodes of hepatic encephalopathy appears to be unrelated to the cause of cirrhosis,increases in the frequency and severity of such episodes predict an increased risk of death.A small metaanalysis determined that lactulose and lactitol were equally effective in the treatment of HE.Probiotics alter the gut flora resulting in decreased ammonia production and absorption due to decreased intraluminal pH. Also shown to alter the short chain fatty acid production, & decrease intestinal permeability.Various studies have shown some improvement in either the prevalence of minimal hepatic encephalopathy or results in neuropsychological tests with the use of probiotics.Lactulose and probiotics improves minimal hepatic encephalopathy in cirrhotic patients and it has also been shown that minimal hepatic encephalopathy predisposes the cirrhotic patient to HE.We will assess the effects of lactulose and probiotics for the prevention of recurrence of hepatic encephalopathy (secondary prophylaxis) in patients after the recovery of an episode of overt hepatic encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis and previous history of recovery from hepatic encephalopathy

Exclusion Criteria:

* history of taking lactulose in the past 6 weeks.
* alcohol intake during the past 6 weeks or during follow up
* patients on secondary prophylaxis for spontaneous bacterial peritonitis
* previous TIPS or shunt surgery
* significant comorbid illness such as heart, respiratory, or renal failure
* any neurologic diseases such as alzheimer's disease, parkinson's disease and nonhepatic metabolic encephalopathies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2008-09; Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
episode of overt hepatic encephalopathy | 6 months

SECONDARY OUTCOMES:
side effects to therapy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Barjesh C Sharma, MD,DM, Principal Investigator — G B Pant Hospital New Delhi 110002
Locations (1):
- G B Pant Hospital, New Delhi, National Capital Territory of Delhi, India